CLINICAL TRIAL: NCT03984383
Title: Regulation of IL33, Endocan and Their Targets in Primary Human Endothelial Cells
Brief Title: IL-33, Endocan and Endothelial Cells
Acronym: IL-33
Status: Withdrawn | Type: Observational
Why Stopped: No extension of ethic comitee
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_13; 2018-A03087-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-05-27; First posted 2019-06-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Endothelial Cell
Keywords: Endothelial cells; inflammation; endothelial dysfunction; IL-33; Endocan
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung-derived endothelial cells: Every patient of more than 18 years undergoing lung cancer surgery in the department of thoracic surgery of the University Hospital of Lille.
- Umbilical cord-derived endothelial cells: Every patient of more than 18 years giving birth in the University Hospital of Lille in the absence of significant materno-foetal disorder (for example: meconium-stained amniotic fluid, chorioamnionitis, placental thrombosis, eclampsia etc.) or of infection for HIV, VHB, VHC or if unknown status for HIV, VHB, VHC the day of the childbirth.

SUMMARY:
The study aims to investigate the inflammatory response of endothelial cells to various stimulations, in particular the production of IL33 and of endocan in response to allergens, agonists of microorganisms and pollutants.

For that purpose, this project attempts to set up a biological collection of lung and umbilical cord endothelial cells.

Lung endothelial cells are resected from a surgical specimen, resulting from a lung cancer surgery.

Umbilical cord-derived endothelial cells are taken from the umbilical cord collected during the delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* signed consent
* Pregnant woman for umbilical cord-derive-endothelial cells

Exclusion Criteria:

* Age < 18 years
* Refusal to participate to the study
* Endothelial cord-drived endothelial cells :

  * significant materno-foetal disorder (for example: meconium-stained amniotic fluid, chorioamnionitis, placental thrombosis, eclampsia etc.)
  * infection for HIV, VHB, VHC
  * unknown status for HIV, VHB, VHC the day of the childbirth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung-derived endothelial cells : every patient of more than 18 years undergoing lung cancer surgery in the department of thoracic surgery of the University Hospital of Lille.
  Umbilical cord-derived endothelial cells : every patient of more than 18 years giving birth in the University Hospital of Lille in the absence of significant materno-foetal disorder (for example: meconium-stained amniotic fluid, chorioamniotis, placental thrombosis, eclampsia etc.) or of infection for HIV, VHB, VHC or if unknown status for HIV, VHB, VHC the day of the childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
change in the level of messenger RNA expressed as IL-33 / GAPDH ratio between stimulated and unstimulated primary human lung endothelial cells. | change from Baseline at 48 hours after stimulation

SECONDARY OUTCOMES:
change in the level of messenger RNA expressed as IL-33 / GAPDH ratio between stimulated and unstimulated primary human lung endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours after stimulation
change in the level of messenger RNA expressed as IL-33 / GAPDH ratio between stimulated and unstimulated primary human umbilical cord-derived endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in IL33 protein concentration between stimulated and unstimulated primary human lung endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in IL33 protein concentration between stimulated and unstimulated primary human umbilical cord-derived endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in the level of messenger RNA expressed as endocan / GAPDH ratio between stimulated and unstimulated primary human lung endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in the level of messenger RNA expressed as endocan / GAPDH ratio between stimulated and unstimulated primary human umbilical cord-derived endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in endocan protein concentration between stimulated and unstimulated primary human lung endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation
change in endocan protein concentration between stimulated and unstimulated primary human umbilical cord-derived endothelial cells. | change from Baseline at 4 hours, 12h ours, 24 hours and 48 hours after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, Principal Investigator — CHU Lille, Service de Pneumologie et Immuno-Allergologie
Locations (1):
- Hop Calmette Chu Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No